CLINICAL TRIAL: NCT04644094
Title: "Surveillance of Postnatal Steroids Effects on Cardiac Function in Extremely Preterm Infants With Evolving BPD: the SPEC Study."
Brief Title: Postnatal Steroids Effects on Cardiac Function in Extremely Preterm
Acronym: SPEC
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Gabriel Altit, Neonatologist, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2021-7305
Record Dates: First submitted 2020-11-09; First posted 2020-11-25 (Actual); Last update posted 2025-06-17 (Actual); Status verified 2025-06

CONDITIONS: Left Ventricular Hypertrophy
Keywords: Lung ultrasound; Echocardiography; Heart rate variability; Left ventricular hypertrophy; Ductus arteriosus; Dexamethasone
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Ductus Arteriosus, Patent

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: Echocardiography (ECHO) and lung ultrasound (LUS) studies before and after Dexamethasone administration — A. Electrocardiographic (ECG) leads will be place in the patient for electrocardiogram (ECG) recordings.
  B. Echocardiography (ECHO) will be performed by an expert member of the Neonatal Echocardiography team C. Heart Rate Variability (HRV): ECG recordings D. Growth trajectory: body weight, length, head circumference, length/weight ratio at 1-, 2-weeks prior treatment, 1-, 2-, 3-, 4-,6-,8-weeks after treatment, at 36-week PMA.

SUMMARY:
Hypothesis/Study question

In infants born at less than 29 weeks of estimated gestational age, what are the effects of dexamethasone use on cardiac structure/performance and lung water content?

Study objectives

To measure effects before and after dexamethasone administration on cardiac structure/performance will be evaluated by using the M-mode technique (Devereux method (25-27) and lung water content will be specifically determined by the degree of water retention in premature lungs assessed by lung ultrasound at the pre specified time points.

Methodology / Study design

Single center, prospective observational cohort study planning to enroll eligible patients over a period of 12 months

DETAILED DESCRIPTION:
This study investigates the effects of dexamethasone on cardiac structure/performance and lung water content in the extremely preterm population undergoing treatment for significant lung disease. For that, the specific aims are to determine the occurrence, evolution over time and possible hemodynamic impact of left ventricular hypertrophy and occurrence and degree of water retention in premature lungs, after dexamethasone administration. As secondary outcomes, this study also investigates the effects of dexamethasone on the ductus arteriosus, body growth, and autonomic regulation heart rate variability, as well as other important outcomes outlined in this protocol.

This study hypothesize that in some infants dexamethasone will be associated with the occurrence of early and/or prolonged left ventricular hypertrophy, which may be associated with changes in cardiac performance. It also hypothesize that the anti-inflammatory effects of dexamethasone would improve inflammation of immature lungs, leading to a decrease in interstitial fluid.

ELIGIBILITY:
Inclusion Criteria:

* < 29 weeks of gestational age at birth admitted at the McGill University Children Hospital's neonatal intensive care unit
* To be initiated on dexamethasone therapy for treatment of significant lung disease as per medical team decision.

Exclusion Criteria:

* Congenital heart disease (except: Atrial septum defect (ASD), Ventricular septum defect (VSD)
* Major congenital anomalies/genetic disorder (Trisomy 13, 18, 21)
* Congenital severe lung or airway malformation (Trachea-esophageal fistula, congenital pulmonary airway malformation, congenital diaphragmatic hernia)
* Twin-twin transfusion syndrome

Min Age: 1 Minute | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Extreme premature babies (< 29 weeks of gestational age at birth) undergoing first treatment with dexamethasone for significant lung disease at the neonatal intensive care.
Sampling Method: Non-Probability Sample
Enrollment: 21 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Left ventricular hypertrophy (LVH) measures by M-mode (Z-Scores) | At the time of echocardiography
  The effects of dexamethasone administration on cardiac structure/performance will be evaluated by using the M-mode technique (Devereux method (25-27)
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
Lung water content | At the time of echocardiography
  Lung water content will be specifically determined by the degree of water retention in premature lungs assessed by lung ultrasound at the specified time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer

SECONDARY OUTCOMES:
Left ventricular (LV) output | At the time of echocardiography
  The effects of dexamethasone administration on:
  On the LV output assessed by Doppler by echocardiography
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
LV and RV function by strain | At the time of echocardiography
  LV and RV function by strain by post treatment of echocardiography acquired images with a Tomtec platform
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
LV ejection fraction | At the time of echocardiography
  The effects of dexamethasone administration on:
  The ejection fraction measured by Simpson on a echocardiography.
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
Ductal size | At the time of echocardiography
  The effects of dexamethasone administration on the size patent ductus arteriosus (PDA) measured on the echocardiography
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
Doppler flow velocities | At the time of echocardiography
  The effects of dexamethasone administration on:
  The Doppler flow velocities measured by echocardiography
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
Measures of PDA significance | At the time of echocardiography
  The effects of dexamethasone administration on:
  LA:AO (left atrium: aorta) Resistance index (RI) of the Anterior Cerebral Artery Direction of ductal flow Peak velocity of PDA in systole
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
LV mass by STE | At the time of echocardiography
  LV mass calculation using Speckle tracking echocardiography (STE) on the Tomtec platform
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
RV function by TAPSE | At the time of echocardiography
  The effects of dexamethasone administration on:
  Tricuspid annular plane systolic excursion measurement by M-Mode on the echocardiography
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
Strain and 3D values | At the time of echocardiography
  The effects of dexamethasone administration on:
  RV and LV strains and on the cardiac volumes by 3 D (RV and LV) by echocardiography acquired images, using Tomtec platform for post treatment
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
Heart rate variability | At the time of echocardiography
  The effects of dexamethasone administration on heart rate variability by ECG
  Time points:
  0 day (before the start of dexamethasone), 3- , 7-day of treatment, 14-day of treatment if still receiving dexamethasone, and 1-week, 2-weeks after dexamethasone discontinuation, and finally at 35 - 37 weeks post menstrual age (PMA) or prior to discharge/transfer
Growth trajectory | At the time of the last echocardiography
  The effects of dexamethasone administration on growth trajectory (body, length, head circumference, L/W ratio) at 1-,2-weekks prior treatment and 1-,2-,3-,4-,6-,8- weeks after treatment, and finally at 36 weeks PMA
Cortisol levels | At the study completion (12 months)
  The effects of dexamethasone after administration:
  Cortisol levels in nmol/L
BPD | At the study completion (12 months)
  The effects of dexamethasone administration on:
  -BPD rate (%) (2018 NICHD definition)
Mortality | At the study completion (12 months)
  - Rate of death in this high risk population (%)
Responders and non responders to Dexamethasone | At the study completion (12 months)
  We will analyze the rate (%) of responders and non-responders to Dexamethasone. Responders: Defined by decreasing Respiratory Severity Scores (RSS) by 40% at day 6 of Dexamethasone treatment or before. RSS is calculated by using maximum of mean airway pressure (MAP) multiplied by fractional oxygen (FiO2) at the day of the first dose of Dexamethasone administration (Day 0)

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Altit, MD, Principal Investigator — Montreal Children's hospital, MUHC
Locations (1):
- Montreal Children's hospital, Mcgill University Health Centre, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No